CLINICAL TRIAL: NCT03571256
Title: A Well-Controlled, Fixed-Dose Study of TEV-50717 (Deutetrabenazine) for the Treatment of Tics Associated With Tourette Syndrome
Brief Title: A Study to Test if TEV-50717 is Effective in Relieving Tics Associated With Tourette Syndrome (TS)
Acronym: ARTISTS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Nuvelution TS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV50717-CNS-30060; 2017-002976-24 (EudraCT Number)
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TEV-50717 High-Dose (Experimental): TEV-50717 tablets twice daily (BID) up to 48 milligrams (mg)/day orally for a total of 8 weeks
  Interventions: Drug: TEV-50717; Drug: Placebo
- TEV-50717 Low-Dose (Experimental): TEV-50717 tablets BID up to 36 mg/day orally for a total of 8 weeks
  Interventions: Drug: TEV-50717; Drug: Placebo
- Placebo (Placebo Comparator): Placebo matched to TEV-50717 for a total of 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-50717 — 6-, 9-, 12-, 15-, and 18 mg oral tablets
  Other Names: AUSTEDO, Deutetrabenazine
  Arms: TEV-50717 High-Dose; TEV-50717 Low-Dose
Drug: Placebo — Placebo matched to TEV-50717 tablets will be taken BID.

SUMMARY:
Standard placebo-controlled, double-blind study design (TEV-50717 [low dose and high dose] vs. placebo in a 1:1:1 ratio) was chosen to determine whether study drug treatment results in a statistically significant effect on the tics in participants with TS.

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs at least 44 pounds (20 kg) at baseline.
* Participant meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5™) diagnostic criteria for TS and, in the opinion of the investigator, participant, and parent/legal guardian, the participant's active tics are causing distress or impairment.
* Participant has a TTS of 20 or higher on the YGTSS at screening and baseline.
* Participant is able to swallow study medication whole.
* -Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has a neurologic disorder other than TS that could obscure the evaluation of tics.
* The participant 's predominant movement disorder is stereotypy (coordinated movements that repeat continually and identically) associated with autism spectrum disorder.
* Participant has clinically significant depression at screening or baseline.
* Participant has a history of suicidal intent or related behaviors within 2 years of screening
* Participant has a history of a previous actual, interrupted, or aborted suicide attempt.
* Participant has a first-degree relative who has completed suicide.
* Participant has a confirmed diagnosis of bipolar disorder, schizophrenia, or another psychotic disorder.
* Participant has received Comprehensive Behavioral Intervention for Tics for TS or Cognitive Behavioral Therapy for obsessive-compulsive disorder (OCD) within 4 weeks of screening.
* Participant has received treatment with deep brain stimulation, transmagnetic stimulation, or transcranial direct current stimulation within 4 weeks of the screening visit for reduction of tics.
* Participant has a history of torsades de pointes, congenital long QT syndrome, bradyarrhythmias, or uncompensated heart failure.
* Participant has participated in an investigational drug or device study and received investigational medicinal product (IMP)/intervention within 30 days or 5 drug half-lives of baseline, whichever is longer.
* Participant is a pregnant or lactating female, or plans to be pregnant during the study.
* -Additional criteria apply, please contact the investigator for more information

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (56):
- United States (19):
  - Teva Investigational Site 060-0160, Gainesville, Florida
  - Teva Investigational Site 060-0166, Gulf Breeze, Florida
  - Teva Investigational Site 060-0161, Miami, Florida
  - Teva Investigational Site 060-0151, Orlando, Florida
  - Teva Investigational Site 060-0153, Orlando, Florida
  - Teva Investigational Site 060-0168, Atlanta, Georgia
  - Teva Investigational Site 060-0155, Chicago, Illinois
  - Teva Investigational Site 060-0164, Chicago, Illinois
  - Teva Investigational Site 060-0152, Indianapolis, Indiana
  - Teva Investigational Site 060-0158, Louisville, Kentucky
  - Teva Investigational Site 060-0167, Rockville, Maryland
  - Teva Investigational Site 060-0165, Ann Arbor, Michigan
  - Teva Investigational Site 060-0170, Bridgeton, Missouri
  - Teva Investigational Site 060-0154, New York, New York
  - Teva Investigational Site 060-0169, Charleston, South Carolina
  - Teva Investigational Site 060-0157, Memphis, Tennessee
  - Teva Investigational Site 060-0156, Nashville, Tennessee
  - Teva Investigational Site 060-0163, Fort Worth, Texas
  - Teva Investigational Site 060-0162, Everett, Washington
- Argentina (5):
  - Teva Investigational Site 060-1407, Buenos Aires
  - Teva Investigational Site 060-1401, Buenos Aires
  - Teva Investigational Site 060-1402, Buenos Aires
  - Teva Investigational Site 060-1403, La Plata
  - Teva Investigational Site 060-1404, Mendoza
- Australia (2):
  - Teva Investigational Site 060-1802, Liverpool
  - Teva Investigational Site 060-1801, Parkville
- Colombia (4):
  - Teva Investigational Site 060-1503, Bello
  - Teva Investigational Site 060-1501, Medellín
  - Teva Investigational Site 060-1506, Medellín
  - Teva Investigational Site 060-1504, Pereira
- Hungary (2):
  - Teva Investigational Site 060-0901, Budapest
  - Teva Investigational Site 060-0902, Szeged
- Italy (4):
  - Teva Investigational Site 060-1005, Cagliari
  - Teva Investigational Site 060-1001, Catania
  - Teva Investigational Site 060-1003, Naples
  - Teva Investigational Site 060-1004, Rome
- Mexico (4):
  - Teva Investigational Site 060-1601, Culiacán
  - Teva Investigational Site 060-1603, León
  - Teva Investigational Site 060-1602, Monterrey
  - Teva Investigational Site 060-1604, Monterrey
- Poland (6):
  - Teva Investigational Site 060-1104, Gdansk
  - Teva Investigational Site 060-1101, Katowice
  - Teva Investigational Site 060-1105, Krakow
  - Teva Investigational Site 060-1102, Poznan
  - Teva Investigational Site 060-1106, Torun
  - Teva Investigational Site 060-1103, Warsaw
- South Korea (4):
  - Teva Investigational Site 060-1901, Seoul
  - Teva Investigational Site 060-1903, Seoul
  - Teva Investigational Site 060-1904, Seoul
  - Teva Investigational Site 060-1902, Seoul
- Ukraine (6):
  - Teva Investigational Site 060-2003, Dnipropetrovsk
  - Teva Investigational Site 060-2001, Kharkiv
  - Teva Investigational Site 060-2002, Kharkiv
  - Teva Investigational Site 060-2007, Kiev
  - Teva Investigational Site 060-2005, Kyiv
  - Teva Investigational Site 060-2006, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Coffey B, Jankovic J, Claassen DO, Jimenez-Shahed J, Gertz BJ, Garofalo EA, Stamler DA, Wieman M, Savola JM, Gordon MF, Alexander JK, Barkay H, Harary E. Efficacy and Safety of Fixed-Dose Deutetrabenazine in Children and Adolescents for Tics Associated With Tourette Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2129397. doi: 10.1001/jamanetworkopen.2021.29397. PMID 34661664

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 158 participants were randomized in a 1:1:1 ratio to TEV-50717 high-dose, TEV-50717 low-dose or placebo group.
Period: Overall Study
Arm/Group | TEV-50717 High-Dose | TEV-50717 Low-Dose | Placebo
Started (Intent-to-treat (ITT) analysis set: all randomized participants) | 52 | 54 | 52
Safety Analysis Set (Received at least 1 dose of study drug) | 52 | 54 | 51
Modified ITT (mITT) Analysis Set (Received at least 1 dose of study drug; had both baseline & at least 1 postbaseline YGTSS assessment) | 49 | 53 | 51
Completed | 46 | 51 | 48
Not Completed | 6 | 3 | 4
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Other than specified | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants.
Groups:
- TEV-50717 High-Dose: TEV-50717 tablets BID up to 48 mg/day orally for a total of 8 weeks
- Total: Total of all reporting groups
Arm/Group | TEV-50717 High-Dose | TEV-50717 Low-Dose | Placebo | Total
Number analyzed (Participants) | 52 | 54 | 52 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (2.63) | 11.7 (2.70) | 11.8 (2.62) | 11.7 (2.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 12 | 39
  Male | 37 | 42 | 40 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 15 | 32
  Not Hispanic or Latino | 43 | 45 | 37 | 125
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 48 | 39 | 135
  Black | 0 | 1 | 0 | 1
  Asian | 0 | 3 | 4 | 7
  Native American | 1 | 1 | 2 | 4
  Multiple | 0 | 0 | 2 | 2
  Other | 3 | 1 | 5 | 9
Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) [Mean (Standard Deviation); unit: units on a scale] — YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 for severe). Motor tic severity score (MTSS) is the sum of 5 items for motor tic severity and vocal tic severity score (VTSS) is the sum of 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome.
  units on a scale | 33.9 (6.17) | 32.9 (7.20) | 34.7 (6.29) | 33.8 (6.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the TTS of the YGTSS at Week 8 Between High-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: YGTSS rating scale is a semi-structured clinician rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic tics. YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 to severe). MTSS is the sum of the 5 items for motor tic severity and VTSS is the sum of the 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome. Least square (LS) mean and standard error (SE) was calculated using mixed-model repeated-measures (MMRM) with treatment group, week (3 levels: Weeks 2, 4, and 8), and the treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6 to 11 years, 12 to 16 years) as covariates.
Time Frame: Baseline, Week 8
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline YGTSS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 High-Dose | Placebo
Number analyzed (Participants) | 49 | 51
units on a scale | -7.8 (1.24) | -7.0 (1.16)
Statistical Analysis 1: Comparison: TEV-50717 High-Dose vs Placebo; Test type: Other; p = 0.600, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -0.8, 95% CI 2-sided [-3.9 to 2.3]

2. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Clinical Global Impression (TS-CGI) Score at Week 8 Between High-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: The TS-CGI scale is a 7-point Likert scale that allows the clinician to use all available information to assess the impact of tics on the participant's quality of life. The TS-CGI is rated as follows: 1 (normal or no tics at all), 2 (borderline), 3 (mild), 4 (moderate), 5 (marked), 6 (severe), and 7 (extreme, incapacitating tics). Lower scores indicate better quality of life. LS mean and SE was calculated using MMRM with treatment group, week (3 levels: Weeks 2, 4, and 8), and the treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6 to 11 years, 12 to 16 years) as covariates.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 High-Dose | Placebo
Number analyzed (Participants) | 49 | 51
units on a scale | -0.8 (0.14) | -0.6 (0.13)

3. Secondary Outcome: Change From Baseline in the TTS of the YGTSS at Week 8 Between Low-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: YGTSS rating scale is a semi-structured clinician rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic tics. YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 to severe). MTSS is the sum of the 5 items for motor tic severity and VTSS is the sum of the 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome. LS mean and SE was calculated using MMRM with treatment group, week (3 levels: Weeks 2, 4, and 8), and the treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6 to 11 years, 12 to 16 years) as covariates.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 53 | 51
units on a scale | -5.9 (1.18) | -7.0 (1.16)

4. Secondary Outcome: Change From Baseline in the TS-CGI Score at Week 8 Between Low-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 53 | 51
units on a scale | -0.6 (0.13) | -0.6 (0.13)

5. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Patient Global Impression of Impact (TS-PGII) Score at Week 8 Between High-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: The TS-PGII is a single-item questionnaire that asks the participant to assess the degree of impact due to current tics (How much do your current tics disrupt things in your life?). The TS-PGII uses a 5-point scale, ranging from not at all (1) to very much (5), to assess overall response to therapy.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 High-Dose | Placebo
Number analyzed (Participants) | 49 | 51
units on a scale | -0.8 (0.17) | -0.7 (0.16)

6. Secondary Outcome: Change From Baseline in the TS-PGII Score at Week 8 Between Low-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 53 | 51
units on a scale | -0.7 (0.15) | -0.7 (0.16)

7. Secondary Outcome: Change From Baseline in the Child and Adolescent Gilles de la Tourette Syndrome - Quality of Life (C&A-GTS-QOL) Activities of Daily Living (ADL) Subscale Score at Week 8 Between High-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: C&A-GTS-QOL is a 27-item questionnaire that asks participant to assess the extent to which their quality of life is impacted by their symptoms. C&A-GTS-QOL contains 6 subscales (cognitive, coprophenomena, psychological, physical, obsessive-compulsive, and ADL) and uses a 5-point Likert scale ranging from no problem to extreme problem. Following 3 questions from 27-item questionnaire were assessed in ADL C&A-GTS-QOL subscale: Question 2 (Had difficulty with school or sport activities?), 24 (Felt you needed more help or support from other people?), and 26 (Had difficulty going out with other people?). Total score of ADL subscale ranged from 0 (no problem) to 12 (extreme problem). Lower score indicated better quality of life. LS mean and SE was calculated using MMRM with treatment group, week (3 levels: Weeks 2, 4, and 8), and treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6-11 years, 12-16 years) as covariates.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 High-Dose | Placebo
Number analyzed (Participants) | 49 | 51
units on a scale | -10.3 (2.85) | -9.0 (2.66)

8. Secondary Outcome: Change From Baseline in the C&A-GTS-QOL ADL Subscale Score at Week 8 Between Low-Dose TEV-50717-Treated Participants and Placebo-Treated Participants
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 53 | 51
units on a scale | -10.0 (2.68) | -9.0 (2.66)

9. Secondary Outcome: Change From Baseline in the Children's Depression Inventory Second Edition (CDI-2; Parent Version and Self-reported Version) Total Score at Week 9
Description: CDI-2 self-report: 28-item questionnaire assessing depressive symptoms in children 7 to 17 years of age with basic reading and comprehension skills. Children were asked to choose 1 of 3 statements that most closely aligns with their feelings in past 2 weeks. It contains 6 subscales (emotional problem, negative mood/physical symptoms, negative self-esteem, functional problems, ineffectiveness, interpersonal problems). Total score: sum of all subscales scores, ranging from 0 to 56, with higher score indicating greater depression severity.CDI-2 parent: 17-item questionnaire administered to parents to assess depression-related behaviors observed in their children. Parents were asked to rate their child's behaviors in past 2 weeks on a 4-point Likert scale from "not at all" to "much or most of the time." It contains 2 subscales (emotional problems and functional problem). Total score: sum of 2 subscales, ranging from 0 to 51, with higher score indicating more depression-related behaviors.
Time Frame: Baseline, Week 9
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717 High-Dose | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 52 | 54 | 51
units on a scale
  CDI-2 Parent Version: number analyzed (Participants) | 45 | 52 | 48
  CDI-2 Parent Version | -1.2 (6.53) | -3.8 (6.34) | -0.8 (5.36)
  CDI-2 Self-Reported Version: number analyzed (Participants) | 45 | 49 | 46
  CDI-2 Self-Reported Version | -2.0 (4.13) | -2.6 (4.90) | -0.4 (4.99)

10. Secondary Outcome: Number of Participants at Baseline and Week 9 With Any Suicidal Ideation or Suicidal Behavior According to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS included responses for Suicidal Ideation or Suicidal Behavior in following 10 categories: 1 = Wish to be dead; 2 = Non-specific active suicidal thoughts; 3 = Active suicidal ideation with any methods (not plan) without intent to act; 4 = Active suicidal ideation with some intent to act, without specific plan; 5 = Active suicidal ideation with specific plan and intent; 6 = Preparatory acts or behavior; 7 = Aborted attempt; 8 = Interrupted attempt; 9 = Non-fatal suicide attempt; and 10 = Completed suicide. Number of participants with any suicidal ideation or suicidal behavior are reported. Any Suicidal ideation or Suicidal Behavior events reported as TEAEs along with all other reported TEAEs are included in the AE module.
Time Frame: Baseline, Week 9
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-50717 High-Dose | TEV-50717 Low-Dose | Placebo
Number analyzed (Participants) | 52 | 54 | 51
Participants
  Baseline | 0 | 0 | 2
  Week 9: number analyzed (Participants) | 46 | 52 | 48
  Week 9 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to follow-up (Week 10)
Description: Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | TEV-50717 High-Dose | TEV-50717 Low-Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 19/52 | 16/54 | 12/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-50717 High-Dose (N=52) | TEV-50717 Low-Dose (N=54) | Placebo (N=51)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-50717 High-Dose (N=52) | TEV-50717 Low-Dose (N=54) | Placebo (N=51)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (5)
Fatigue (General disorders) | 5 (6) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 2 (2) | 3 (4)
Increased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 6 (8) | 8 (13) | 4 (4)
Somnolence (Nervous system disorders) | 8 (11) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03571256/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03571256/SAP_001.pdf